CLINICAL TRIAL: NCT00541320
Title: Dose Ranging Trial for the Evaluation of the Safety and Efficacy of GW813893 in the Prophylaxis of Venous Thromboembolism Post Total Knee Replacement Surgery.
Brief Title: Phase IIa Venous Thromboembolism (VTE) Prevention Study In Total Knee Replacement (TKR)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No longer viable
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FTI102595
Record Dates: First submitted 2007-02-12; First posted 2007-10-10 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Venous Thromboembolism
Keywords: Anti-thrombolytic direct Factor Xa inhibitor
MeSH Terms: conditions — Venous Thromboembolism | interventions — 2-(5-chlorothien-2-yl)-N-(1-(1-methyl-2-(morpholin-4-yl)-2-oxoethyl)-2-oxopyrrolidin-3-yl)ethenesulfonamide

INTERVENTIONS:
Drug: GW813893

SUMMARY:
This study was designed to assess the safety and efficacy of GW813893 in the prophylaxis of VTE following TKR and to provide evidence to enable the selection of the appropriate dose(s) and dose regimen of GW813893 for future investigation.

ELIGIBILITY:
Inclusion criteria:

* Patients who are scheduled for primary elective unilateral total knee arthroplasty.

Exclusion criteria:

* Women who are not surgically sterile or post-menopausal
* Have a contra-indication to contract venography
* Have a known disorder associated with increased risk of bleeding or have been immobile up to 12 weeks before surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Incidence of death OR symptomatic or non-symptomatic blood clots in the legs OR symptomatic blood clots in the lungs within 7 +/- 2 days following total knee replacement surgery. | symptomatic blood clots in the lungs within 7 +/- 2 days following total knee replacement surgery.

SECONDARY OUTCOMES:
Incidence of bleeding within 7 +/- 2 days following total knee replacement surgery. | Incidence of bleeding within 7 +/- 2 days following total knee replacement surgery

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (8):
- United States (8):
  - GSK Clinical Trials Call Center, Birmingham, Alabama
  - GSK Clinical Trials Call Center', Phoenix, Arizona
  - GSK Clinical Trials Call Center, Phoenix, Arizona
  - GSK Clinical Trials Call Center, Yuba City, California
  - GSK Clinical Trials Call Center, St. Petersburg, Florida
  - GSK Clinical Trials Call Center, Decatur, Georgia
  - GSK Clinical Trials Call Center, Charleston, South Carolina
  - GSK Clinical Trials Call Center, San Antonio, Texas